CLINICAL TRIAL: NCT01283646
Title: Multicenter Clinical Study, Phase III, Randomized, Double-blind, of Prospectively Evaluate the Effectiveness and Tolerability of Apevitin BC Comparing to Vitamin Complex in Appetite Stimulation
Brief Title: Efficacy and Tolerability of Apevitin BC Comparing to Vitamin Complex in Stimulating the Appetite
Acronym: Inappetence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRPEMS0910
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2013-03

CONDITIONS: Lack or Loss Appetite Nonorganic Origin
MeSH Terms: interventions — Vitamin B Complex; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apevitin BC (Experimental): Children (5 to 6 years): 3.5 ml 3 times a daily Children (7 to 15 years): 5 ml 3 times a daily
  Interventions: Drug: Apevitin BC
- Vitamin B Complex + Vitamin C (Active Comparator): Children (5 to 6 years): 3.5 ml 3 times a daily Children (7 to 15 years): 5 ml 3 times a daily
  Interventions: Drug: Vitamin B Complex + Vitamin C

INTERVENTIONS:
Drug: Apevitin BC — 3.5 to 5 ml 3 times a daily
  Arms: Apevitin BC
Drug: Vitamin B Complex + Vitamin C — 3.5 to 5 ml 3 times a daily
  Arms: Vitamin B Complex + Vitamin C

SUMMARY:
Lack of appetite is one of the most common reasons for visits to pediatric clinics.The symptoms usually manifest after weaning when they are introduced into the diet of infant foods containing salt.Is normally used to cyproheptadine in conjunction with vitamins C and B and also vitamins complex.

DETAILED DESCRIPTION:
Study Design:

* Multicenter
* Phase III
* Randomized
* Double Blind
* Prospective and Comparative
* Experiment duration: 30 days
* 3 visits (day 0, day 15 and day 30)
* Increased appetite
* Adverse event

ELIGIBILITY:
Inclusion Criteria:

* Patients with inappetence;
* Wash out 20 days after ingestion before similar drug;
* The charge of the patient must understand and consent in writing;
* Responsible for the minor must be able to understand the study procedures, agree to participate and give written consent.

Exclusion Criteria:

* Patients with intestinal parasitoses infection;
* Patients with glaucoma open or closure angle;
* Patients with predisposition to urinary retention;
* Patients with stenosis peptic ulcer or pylorus - duodenal obstruction;
* Debilitated patients or in acute attack of asthma;
* Patients who have lass of appetite caused by any serious disease;
* Patients who make use of any drugs central nervous system depressants;
* Patients who make use of medicines monoamineoxidase inhibitors, tricyclic antidepressants, phenothiazines, probenecid, levodopa, phenytoin, Phenobarbital, chloramphenicol, cyclosphosphamide, cyclosporine, chlorambucil,corticotropin, mercaptopurine, isoniazid , penicillin, estrogens, contraceptives, haloperidol, ipratropium, barbiturates, primidone, salicylates.
* Hypersensitivity to components of the formula
* Patients who is participating in another clinical study;
* No able to adhere to protocol;
* Any pathology or past medical condition that can interfere with this protocol.
* Other conditions deemed reasonable by the medical investigator as to the disqualification of the individual from study participation.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of Apevitin BC in appetite stimulation compared to vitamin complex. | 30 days
  Clinical evaluation of the patient's general condition. The lowest responsible will report less data about their inappetence.

SECONDARY OUTCOMES:
Evaluate the tolerability of Apevitin BC in stimulating the appetite compared to vitamin complex | 30 days
  The lowest responsible will repost less data about their inappetence.Final evaluation of efficacy and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Pinho, MD, Study Director — EMS
Locations (3):
- Brazil (3):
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Clínica A/Z, São Paulo, São Paulo
  - Clínica Dr. Felício Savioli, São Paulo, São Paulo